CLINICAL TRIAL: NCT07271290
Title: Preventing Noise Exposure in Farmworkers
Acronym: POP
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Laura Coco, Assistant Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-25-0158; 1K23DC022303-01A1 (NIH)
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Noise Exposure
Keywords: noise exposure; hearing loss; farmworker
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Multilevel Intervention Group) (Experimental): This group will receive a multilevel intervention designed to reduce occupational noise exposure on farms. The intervention includes the following components:
  Farmworker-level strategies: Provision of earplugs and brief training on hearing protection and noise risks.
  Supervisor/manager training: Short training sessions for supervisors on the importance of noise control and how to support hearing conservation on the farm.
  Environmental modifications: Placement of signs and earplug dispensers at high-noise areas throughout the farm.
  The intervention will be implemented over a short time frame, and noise exposure will be measured before and one month after the intervention.
  Interventions: Behavioral: Protected Ears Project
- Control Arm (Usual Practice) (No Intervention): Farms in the control group will not receive any intervention during the study period. Farmworkers on these farms will participate in baseline and follow-up data collection but will not receive hearing protection materials, training, or signage during the trial.
  These farms will be offered the intervention after study completion, pending feasibility and interest.

INTERVENTIONS:
Behavioral: Protected Ears Project — This multilevel intervention is specifically designed for agricultural worksites and targets noise exposure reduction among farmworkers. Unlike standard educational or PPE-only approaches, this intervention integrates behavioral, supervisory, and environmental strategies across three levels:
  Farmworkers receive training and are provided with earplugs along with visual demonstrations on correct use.
  Supervisors/managers participate in brief training that emphasizes their role in promoting hearing protection and supporting safe practices.
  Environmental modifications include installing signage in high-noise areas and accessible earplug dispensers at strategic locations across the farm.
  This integrated approach is tailored to the unique language, literacy, and occupational context of farmworkers in the US southwest region. It is also designed for feasibility and scalability in real-world agricultural settings.
  Arms: Intervention Arm (Multilevel Intervention Group)

SUMMARY:
This study will evaluate a multilevel intervention designed to reduce hazardous noise exposure among farmworkers. The intervention includes training for farmworkers and supervisors, placement of safety signage, and distribution of hearing protection at noisy worksites.

The research has two primary goals: (1) to determine whether the intervention decreases the amount of time farmworkers are exposed to hazardous noise, and (2) to identify barriers and facilitators to implementing the intervention in agricultural settings.

The study includes two parts. In Part I, a small group of farmworkers will participate in an adapted hearing-protection training and complete pre- and post-training assessments of earplug fit, knowledge, attitudes, and behaviors. In Part II, farmworkers will wear personal sound level meters before and after the intervention to measure changes in noise exposure, and both farmworkers and supervisors will complete surveys about perceptions of noise and intervention components. Some participants may also be invited to complete interviews about their experiences.

Results will inform refinement and scale-up of the intervention to support hearing-loss prevention in agricultural workplaces.

DETAILED DESCRIPTION:
Noise-induced hearing loss (NIHL) is a preventable occupational condition, yet farmworkers are routinely exposed to hazardous noise and rarely use hearing protection. This study will evaluate a multilevel intervention designed to improve hearing-protection practices in agricultural settings. The intervention includes (1) a culturally tailored training for farmworkers, (2) a complementary training for supervisors, (3) safety signage placed in high-noise areas, and (4) distribution of foam earplugs at designated work locations.

Part I (Farmworker-Level Training Evaluation)

A group of farmworkers (n ≈ 15) will complete pre-training assessments, including baseline fit testing of foam earplugs using a standardized Personal Attenuation Rating (PAR) device. Participants will then view an adapted, Spanish-language digital training module that includes information on NIHL risks and step-by-step instruction on proper earplug insertion. After viewing the module, participants will complete post-training PAR testing, as well as a brief survey assessing knowledge, attitudes, and behaviors related to hearing protection. Open-ended questions will capture immediate reactions and perceived usefulness of the training.

Part II (Multilevel Intervention Evaluation)

Following the training, the full multilevel intervention will be implemented at participating farms. Farmworkers will wear personal sound level meters before and after the intervention period to capture changes in noise exposure. Surveys administered to farmworkers and supervisors will measure perceptions of noise hazards, use of hearing protection, and impressions of the intervention components. A subset of participants may be invited to complete semi-structured interviews to identify barriers and facilitators to implementing the intervention under typical agricultural working conditions.

Outcomes and Use of Results

Primary outcomes include changes in hazardous noise exposure and feasibility of implementing the multilevel intervention on farms. Secondary outcomes include improvements in earplug fit (PAR), knowledge and attitudes related to hearing protection, and participant-reported acceptability and appropriateness of the intervention.

Findings will support refinement of the intervention and inform a future larger-scale study aimed at preventing noise-induced hearing loss among agricultural workers.

ELIGIBILITY:
Inclusion Criteria:

* Farmworkers and supervisors

Exclusion Criteria:

* Not a farmworker or supervisor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Noise exposure | baseline and 1 month post intervention
  Noise exposure levels (8-hr time-weighted average decibel level, accounting for hearing protection).

IPD SHARING:
Plan to Share IPD: Undecided